CLINICAL TRIAL: NCT05158660
Title: Assessment of Intracerebral Hematoma Using Transcranial Duplex _ Hospital Based Study
Brief Title: Assessment of Intracerebral Hematoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Mohammed Gafar, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: intracerebral hematoma
Record Dates: First submitted 2021-12-03; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Intracerebral Hematoma
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients assessed by transcranial duplex sonography (Experimental)
  Interventions: Device: transcranial duplex sonography

INTERVENTIONS:
Device: transcranial duplex sonography — it is an imaging device that will measure the intracerebral hematoma expansion

SUMMARY:
The study will assess acute intracerebral hematoma expansion within the first 48 hours from the onset using transcranial duplex sonography in patients who have acute intracerebral hematoma , and will also assess the correlation between the transcranial duplex sonography measurements and the clinical outcome of these patients .

ELIGIBILITY:
Inclusion Criteria:

1. first ever non traumatic supratentorial primary intracerebral haemorrhage on non contrast CT brain
2. admitted within 24 hours of symptom onset

Exclusion Criteria:

1. blood diseases, decompansated hepatic or renal impairment, or encephalopathy caused by electrolyte disturbance
2. on anticoagulant treatment
3. if devolped major complications during hospitalization ( e.g sever chest infection, hypoxia, or deep venous thrombosis )
4. comorbid neurological or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
change from baseline in volume of intracerebral hematoma | at baseline, then 24 hour after the baseline, and finally 48 hours after the baseline